CLINICAL TRIAL: NCT03655899
Title: Metabolomic Alterations in the Vascular Compartment in Patients With Sepsis - an Observational Study
Brief Title: Metabolomic Alterations in the Vascular Compartment in Patients With Sepsis
Acronym: METSEP
Status: Terminated | Type: Observational
Why Stopped: Analysis of cell phenotypes was not possible
Sponsor: Pär Johansson (Other)
Responsible Party: Sponsor-Investigator, Pär Johansson, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: Metabolomics 16024946
Record Dates: First submitted 2017-09-26; First posted 2018-08-31 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Endothelial Dysfunction
Keywords: metabolomics; systems biology; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Red blood cells, white blood cells, platelets, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the metabolic alterations of vascular cells caused by sepsis and septic shock

DETAILED DESCRIPTION:
This study will investigate the metabolic alterations of vascular cells caused by sepsis and septic shock in 60 patients

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* Sepsis or Septic shock

Exclusion Criteria:

* Pregnant or breastfeeding
* Hemoglobin ≤ 5.0 mmol/L
* Platelets ≤ 5.0 mia/L
* Consent not obtainable
* Do not resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Shock induced endotheliopaty | Up to 30 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Pär Johansson, Study Director — Rigshospitalet, Dept. of Clinical Immunology
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark